CLINICAL TRIAL: NCT02561962
Title: A Phase 1 First in Human Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 224 in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Phase 1 Study in Subjects With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20130314
Record Dates: First submitted 2015-09-25; First posted 2015-09-28 (Estimated); Results first posted 2021-10-07 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Dose Exploration: AMG 224 Dose A (Experimental): Participants were administered AMG 224 Dose A as an intravenous (IV) infusion once every 3 weeks (Q3W) on Day 1 of each cycle, where each cycle is 3 weeks.
  Interventions: Drug: AMG 224
- Dose Exploration: AMG 224 Dose B (Experimental): Participants were administered AMG 224 Dose B as an IV infusion Q3W on Day 1 of each cycle, where each cycle is 3 weeks.
  Interventions: Drug: AMG 224
- Dose Exploration: AMG 224 Dose C (Experimental): Participants were administered AMG 224 Dose C as an IV infusion Q3W on Day 1 of each cycle, where each cycle is 3 weeks.
  Interventions: Drug: AMG 224
- Dose Exploration: AMG 224 Dose D (Experimental): Participants were administered AMG 224 Dose D as an IV infusion Q3W on Day 1 of each cycle, where each cycle is 3 weeks.
  Interventions: Drug: AMG 224
- Dose Exploration: AMG 224 Dose E (Experimental): Participants were administered AMG 224 Dose E as an IV infusion Q3W on Day 1 of each cycle, where each cycle is 3 weeks.
  Interventions: Drug: AMG 224
- Dose Exploration: AMG 224 Dose F (Experimental): Participants were administered AMG 224 Dose F as an IV infusion Q3W on Day 1 of each cycle, where each cycle is 3 weeks.
  Interventions: Drug: AMG 224
- Dose Exploration: AMG 224 Dose G (Experimental): Participants were administered AMG 224 Dose G as an IV infusion Q3W on Day 1 of each cycle, where each cycle is 3 weeks.
  Interventions: Drug: AMG 224
- Dose Expansion: AMG 224 Dose H + prior CD38 targeting antibody treatment (Experimental): Participants who had prior treatment with CD38-targeting antibody were administered AMG 224 Dose H (the maximum tolerated dose [MTD] based on the dose exploration phase) as an IV infusion Q3W on Day 1 of each cycle, where each cycle is 3 weeks.
  Interventions: Drug: AMG 224
- Dose Expansion: AMG 224 Dose H + no prior CD38 targeting antibody treatment (Experimental): Participants who had no prior treatment with CD38-targeting antibody were administered AMG 224 Dose H (the MTD based on the dose exploration phase) as an IV infusion Q3W on Day 1 of each cycle, where each cycle is 3 weeks.
  Interventions: Drug: AMG 224

INTERVENTIONS:
Drug: AMG 224 — Administered as an IV infusion.

SUMMARY:
This is a first in human phase 1 multicenter open label study in subjects with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
This is a first in human phase 1 multicenter open label study to evaluate the safety and tolerability of AMG 224 in subjects with relapsed or refractory multiple myeloma. The study will be conducted in 2 parts. Part 1 is the dose-exploration and part 2 is the dose-expansion. Study medication will be administered once every 3 weeks by intravenous (IV) infusion.

ELIGIBILITY:
Inclusion Criteria:

- Pathologically documented,multiple myeloma relapsed or refractory progressive disease after at least 3 lines of therapy for multiple myeloma.

Prior therapeutic treatment or regimens must include proteasome inhibitors (e.g. bortezomib) and immunomodulatory drugs (e.g. lenalidomide).

* Willing and able to undergo bone marrow aspirate per protocol (with or without bone marrow biopsy per institutional guidelines).
* Measurable disease per the International Myeloma Working Group (IMWG) response criteria
* Hematological function, as follows, without transfusion support:
* Absolute neutrophil count ≥ 1.0 X 10^9/L,
* Platelet count ≥ 75 X 10^9/L (in patients with < 50% of bone marrow nucleated cells were plasma cells) or ≥ 50 X 10^9/L (in patients with ≥ 50% of bone marrow nucleated cells were plasma cells) without transfusion or growth factor support
* Hemoglobin > 8 g/dL (> 80 g/L)
* Adequate renal and hepatic function
* Left ventricular ejection fraction (LVEF) > 50%

Exclusion Criteria:

* Currently receiving treatment in another investigational device or drug study, or less than 28 days since ending treatment on another investigational device or drug study
* Autologous stem cell transplant less than 90 days prior to study day 1
* Multiple myeloma with IgM subtype
* POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) syndrome, Plasma cell leukemia, Waldenstrom's macroglobulinemia or Amyloidosis
* Glucocorticoid therapy (prednisone > 30 mg/day or equivalent) within 7 days prior to study day
* Myocardial infarction within 6 months of study day 1, symptomatic congestive heart failure (New York Heart Association > class II)
* A baseline ECG QTcF > 470 msec
* Anti-tumor therapy (chemotherapy, antibody therapy, molecular targeted therapy, or investigational agent) within 28 days prior to study day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (5):
- United States (4):
  - Research Site, West Hollywood, California
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research Site, Houston, Texas
- Research Site, Prahran, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Lee HC, Raje NS, Landgren O, Upreti VV, Wang J, Avilion AA, Hu X, Rasmussen E, Ngarmchamnanrith G, Fujii H, Spencer A. Phase 1 study of the anti-BCMA antibody-drug conjugate AMG 224 in patients with relapsed/refractory multiple myeloma. Leukemia. 2021 Jan;35(1):255-258. doi: 10.1038/s41375-020-0834-9. Epub 2020 Apr 21. No abstract available. PMID 32317775
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 42 participants were enrolled in the study at 4 research centers in Australia and the United States from 20 November 2015 to 21 April 2022. Primary completion date: 30 Nov 2018.
Pre-assignment Details: Doses of AMG 224 in dose exploration part range from lowest in Dose A (30mg) up to highest in Dose G (250mg). Specific doses are blinded due to the protection of propriety information.
Groups:
- Dose Expansion: AMG 224 Dose H + Prior CD38 Targeting Antibody Treatment: Participants who had prior treatment with CD38-targeting antibody were administered AMG 224 Dose H (the maximum tolerated dose [MTD] identified based on the dose exploration phase) as an IV infusion Q3W on Day 1 of each cycle, where each cycle is 3 weeks.
- Dose Expansion: AMG 224 Dose H + no Prior CD38 Targeting Antibody Treatment: Participants who had no prior treatment with CD38-targeting antibody were administered AMG 224 Dose H (the MTD identified based on the dose exploration phase) as an IV infusion Q3W on Day 1 of each cycle, where each cycle is 3 weeks.
Period: Overall Study
Arm/Group | Dose Exploration: AMG 224 Dose A | Dose Exploration: AMG 224 Dose B | Dose Exploration: AMG 224 Dose C | Dose Exploration: AMG 224 Dose D | Dose Exploration: AMG 224 Dose E | Dose Exploration: AMG 224 Dose F | Dose Exploration: AMG 224 Dose G | Dose Expansion: AMG 224 Dose H + Prior CD38 Targeting Antibody Treatment | Dose Expansion: AMG 224 Dose H + no Prior CD38 Targeting Antibody Treatment
Started | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 11 | 2
Received Treatment | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 9 | 2
Completed | 2 | 3 | 3 | 3 | 4 | 3 | 3 | 7 | 2
Not Completed | 1 | 0 | 0 | 0 | 2 | 3 | 2 | 4 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0
Not completed — Decision by sponsor | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set: all participants that are enrolled and received at least 1 dose of AMG 224.
Groups:
- Dose Exploration: AMG 224 Dose G: Participants were administered AMG 224 Dose G as an intravenous (IV) infusion once every 3 weeks (Q3W) on Day 1 of each cycle, where each cycle is 3 weeks.
- Total: Total of all reporting groups
Arm/Group | Dose Exploration: AMG 224 Dose A | Dose Exploration: AMG 224 Dose B | Dose Exploration: AMG 224 Dose C | Dose Exploration: AMG 224 Dose D | Dose Exploration: AMG 224 Dose E | Dose Exploration: AMG 224 Dose F | Dose Exploration: AMG 224 Dose G | Dose Expansion: AMG 224 Dose H + Prior CD38 Targeting Antibody Treatment | Dose Expansion: AMG 224 Dose H + no Prior CD38 Targeting Antibody Treatment | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 9 | 2 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (7.0) | 63.7 (3.8) | 64.3 (11.2) | 70.7 (4.0) | 60.5 (7.1) | 65.0 (5.7) | 58.2 (6.0) | 71.3 (8.7) | 53.0 (9.9) | 64.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 1 | 3 | 4 | 4 | 4 | 1 | 21
  Male | 2 | 1 | 2 | 2 | 3 | 2 | 1 | 5 | 1 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1 | 1 | 8
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 4 | 4 | 3 | 8 | 1 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black (or African American) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 6
  White | 0 | 1 | 2 | 3 | 4 | 3 | 3 | 7 | 2 | 25
  Other | 3 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose-Limiting Toxicity (DLT)
Description: Adverse events, including DLTs, were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. A DLT was considered as any of the below, if judged by the investigator to be possibly related to AMG 224:
  Hematological:
  * Grade 4 neutropenia lasting > 7 days
  * Grade 3 or 4 neutropenia with fever > 38.5°C
  * Grade 3 thrombocytopenia with ≥ Grade 2 hemorrhage
  * Grade 4 thrombocytopenia lasting > 7 days
  * Grade 3 anemia with symptoms or required intervention
  * Grade 4 anemia
  * Lymphopenia is not considered a DLT
  Non-hematological:
  * ≥ Grade 3 nausea, vomiting or diarrhea persisting > 3 days despite optimal medical support
  * Grade 3 fatigue persisting > 7 days
  * ≥ Grade 3 acute kidney injury lasting > 3 days
  * Elevation of aspartate aminotransferase or alanine aminotransferase >3x to >8x upper limit of normal (ULT) dependent on criteria
  * Total bilirubin > 3x ULN
  Participants meeting the criteria for Hy's Law case were considered to have a DLT.
Time Frame: Day 1 to Day 28
Population: DLT analysis set: all participants who are DLT evaluable. A participant was not DLT-evaluable if the participant discontinued treatment for any reason other than a DLT prior to completing the first 28 days of AMG 224 treatment or did not receive 2 doses of AMG 224 during the 28-day DLT window.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Exploration: AMG 224 Dose A | Dose Exploration: AMG 224 Dose B | Dose Exploration: AMG 224 Dose C | Dose Exploration: AMG 224 Dose D | Dose Exploration: AMG 224 Dose E | Dose Exploration: AMG 224 Dose F | Dose Exploration: AMG 224 Dose G | Dose Expansion: AMG 224 Dose H + Prior CD38 Targeting Antibody Treatment | Dose Expansion: AMG 224 Dose H + no Prior CD38 Targeting Antibody Treatment
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 4 | 8 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0

2. Primary Outcome: Number of Participants With a Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial participant.
  TEAEs were any AE that occurred after receiving at least 1 dose of treatment.
  Treatment-related TEAEs were those considered related to study treatment by the investigator.
  Any clinically significant changes in ECGs, vital signs, physical examination with a neurologic assessment and clinical laboratory tests were recorded as TEAEs.
Time Frame: Day 1 of Cycle 1 to up to the end of Cycle 4, where each cycle is 3 weeks; up to 12 weeks.
Population: Safety analysis set: all participants that are enrolled and received at least 1 dose of AMG 224.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Exploration: AMG 224 Dose A | Dose Exploration: AMG 224 Dose B | Dose Exploration: AMG 224 Dose C | Dose Exploration: AMG 224 Dose D | Dose Exploration: AMG 224 Dose E | Dose Exploration: AMG 224 Dose F | Dose Exploration: AMG 224 Dose G | Dose Expansion: AMG 224 Dose H + Prior CD38 Targeting Antibody Treatment | Dose Expansion: AMG 224 Dose H + no Prior CD38 Targeting Antibody Treatment
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 9 | 2
Participants
  TEAE | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 9 | 2
  Treatment-related TEAE | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 7 | 1

3. Secondary Outcome: Maximum Observed Concentration (Cmax) of AMG 224 Conjugated Antibody, Total Anti-B-cell Maturation Antigen (Anti-BCMA) Antibody, and Total Unconjugated DM1
Description: Cmax of AMG 224 conjugated antibody, total anti-BCMA antibody and total unconjugated DM1 was measured. DM1 is a semi-synthetic derivative of the ansamycin antibiotic, maytansine conjugated to the non-cleavable linker 4-[N-maleimidomethyl] cyclohexane-1-carboxylate conjugated to lysine residues in the antibody (MCC).
Time Frame: AMG 224 and anti-BCMA antibody: pre-dose, 0.5 hours, end of infusion (EOI), 4 hours, 24 hours, 96 hours, 168 hours, and 336 hours post-dose (Cycles 1 + 2); DM1: pre-dose, 0.5 hours, EOI, 4 hours, 24 hours, and 96 hours post-dose (Cycles 1 + 2)
Population: The pharmacokinetic (PK) parameter analysis set included participants who received at least 1 dose of AMG 224 and for whom PK parameters could be adequately estimated.
Measure: Mean (Full Range); unit: µg/mL
Groups:
- Dose Expansion: AMG 224 3 mg/kg: All participants in Dose Expansion who had prior treatment or no prior treatment with a CD38-targeting antibody were administered the MTD of AMG 224 identified in the dose escalation as 3 mg/kg. AMG 224 was administered as an intravenous (IV) infusion once every 3 weeks (Q3W) on Day 1 of each cycle, where each cycle is 3 weeks.
Arm/Group | Dose Exploration: AMG 224 Dose A | Dose Exploration: AMG 224 Dose B | Dose Exploration: AMG 224 Dose C | Dose Exploration: AMG 224 Dose D | Dose Exploration: AMG 224 Dose E | Dose Exploration: AMG 224 Dose F | Dose Exploration: AMG 224 Dose G | Dose Expansion: AMG 224 3 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 6 | 5 | 10
µg/mL
  AMG 224 Conjugated Antibody after Cycle 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 10
  AMG 224 Conjugated Antibody after Cycle 1 | 11.4 [5.99 to 14.3] | 22.0 [16.4 to 28.9] | 25.3 [20.0 to 31.2] | 32.9 [19.8 to 42.9] | 37.5 [6.32 to 67.7] | 54.2 [45.1 to 74.4] | 61.9 [47.1 to 75.5] | 55.8 [39.9 to 80.9]
  AMG 224 Conjugated Antibody after Cycle 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 2 | 8
  AMG 224 Conjugated Antibody after Cycle 2 | 11.5 [8.26 to 15.4] | 29.3 [20.6 to 44.6] | 31.0 [26.4 to 39.0] | 38.5 [24.0 to 51.5] | 40.1 [29.0 to 53.8] | 60.8 [51.2 to 84.7] | 78.7 [67.4 to 89.9] | 73.3 [46.6 to 89.9]
  Total Anti-BCMA Antibody after Cycle 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 10
  Total Anti-BCMA Antibody after Cycle 1 | 11.9 [7.09 to 14.5] | 23.9 [20.4 to 30.5] | 25.3 [21.4 to 29.8] | 34.7 [19.3 to 47.2] | 40.2 [8.72 to 75.8] | 52.4 [49.6 to 55.5] | 67.7 [50.4 to 84.9] | 52.1 [33.7 to 73.8]
  Total Anti-BCMA Antibody after Cycle 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 2 | 8
  Total Anti-BCMA Antibody after Cycle 2 | 11.9 [9.84 to 13.5] | 34.6 [22.5 to 51.8] | 33.2 [28.9 to 40.5] | 41.6 [25.0 to 56.2] | 45.3 [34.6 to 63.9] | 63.4 [55.5 to 72.4] | 79.6 [50.2 to 109] | 62.4 [39.0 to 77.2]
  DM1 after Cycle 1 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.000312 [0.00 to 0.000501] | 0.000549 [0.000445 to 0.000693] | 0.00131 [0.000568 to 0.00210] | 0.00141 [0.000967 to 0.00192] | 0.00155 [0.00123 to 0.00201] | 0.00149 [0.000924 to 0.00210]
  DM1 after Cycle 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 2 | 8
  DM1 after Cycle 2 | 0.00 [0.00 to 0.00] | 0.000119 [0.00 to 0.000356] | 0.000414 [0.000297 to 0.000590] | 0.000654 [0.000423 to 0.000913] | 0.000872 [0.000658 to 0.00121] | 0.00172 [0.00141 to 0.00264] | 0.00161 [0.00151 to 0.00170] | 0.00177 [0.00140 to 0.00242]

4. Secondary Outcome: Minimum Observed Concentration (Cmin) of AMG 224 Conjugated Antibody, Total Anti-BCMA Antibody, and Total Unconjugated DM1
Description: Cmin of AMG 224 conjugated antibody, total anti-BCMA antibody and total unconjugated DM1 was measured.
Time Frame: AMG 224 and anti-BCMA antibody: pre-dose, 0.5 hours, EOI, 4 hours, 24 hours, 96 hours, 168 hours, and 336 hours post-dose (Cycles 1 + 2); DM1: pre-dose, 0.5 hours, EOI, 4 hours, 24 hours, and 96 hours post-dose (Cycles 1 + 2)
Population: The PK parameter analysis set included participants who received at least 1 dose of AMG 224 and for whom PK parameters could be adequately estimated.
Measure: Mean (Full Range); unit: µg/mL
Arm/Group | Dose Exploration: AMG 224 Dose A | Dose Exploration: AMG 224 Dose B | Dose Exploration: AMG 224 Dose C | Dose Exploration: AMG 224 Dose D | Dose Exploration: AMG 224 Dose E | Dose Exploration: AMG 224 Dose F | Dose Exploration: AMG 224 Dose G | Dose Expansion: AMG 224 3 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 6 | 5 | 10
µg/mL
  AMG 224 Conjugated Antibody after Cycle 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 2 | 8
  AMG 224 Conjugated Antibody after Cycle 1 | 1.45 [0.970 to 1.71] | 2.81 [2.11 to 4.05] | 4.54 [3.70 to 5.46] | 4.40 [1.69 to 8.80] | 3.51 [2.11 to 6.32] | 10.5 [5.75 to 18.2] | 9.29 [3.87 to 14.7] | 10.6 [3.65 to 16.6]
  AMG 224 Conjugated Antibody after Cycle 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 2 | 8
  AMG 224 Conjugated Antibody after Cycle 2 | 1.51 [0.811 to 1.93] | 3.06 [2.44 to 4.05] | 6.71 [5.97 to 7.99] | 5.91 [3.33 to 10.1] | 6.64 [1.91 to 12.0] | 15.2 [5.75 to 20.4] | 20.0 [3.87 to 36.2] | 15.9 [4.68 to 27.7]
  Total Anti-BCMA Antibody after Cycle 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 2 | 8
  Total Anti-BCMA Antibody after Cycle 1 | 1.70 [1.05 to 2.07] | 3.91 [2.56 to 5.83] | 6.69 [5.52 to 8.27] | 5.50 [2.78 to 9.87] | 4.86 [2.86 to 8.72] | 13.5 [8.14 to 17.5] | 10.9 [3.47 to 18.3] | 9.47 [3.76 to 15.1]
  Total Anti-BCMA Antibody after Cycle 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 2 | 8
  Total Anti-BCMA Antibody after Cycle 2 | 2.25 [1.25 to 2.78] | 4.62 [3.78 to 5.83] | 11.9 [10.2 to 14.7] | 10.1 [4.24 to 19.1] | 11.3 [3.72 to 21.0] | 21.8 [8.14 to 33.6] | 15.4 [3.47 to 27.4] | 13.1 [4.56 to 23.7]
  DM1 after Cycle 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 6 | 5 | 10
  DM1 after Cycle 1 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.000160 [0.00 to 0.000341] | 0.000268 [0.00 to 0.000353] | 0.000206 [0.00 to 0.000408] | 0.000189 [0.00 to 0.000694]
  DM1 after Cycle 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 5 | 2 | 8
  DM1 after Cycle 2 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.000150 [0.00 to 0.000300] | 0.000468 [0.000443 to 0.000535] | 0.000254 [0.00 to 0.000507] | 0.000494 [0.000364 to 0.000796]

5. Secondary Outcome: Area Under the Concentration-time Curve (AUC) of AMG 224 Conjugated Antibody, Total Anti-BCMA Antibody, and Total Unconjugated DM1
Description: AUC from time zero to 3 weeks (AUC(3 weeks)) was determined for AMG 224 conjugated antibody and total anti-BCMA antibody, and AUC from time zero to 96 hours (AUC(0-96hr)) was determined for DM1.
Time Frame: AMG 224 and anti-BCMA antibody: pre-dose, 0.5 hours, EOI, 4 hours, 24 hours, 96 hours, 168 hours, and 336 hours post-dose (Cycle 1 + 2); DM1: pre-dose, 0.5 hours, EOI, 4 hours, 24 hours, and 96 hours post-dose (Cycles 1 + 2)
Population: The PK parameter analysis set included participants who received at least 1 dose of AMG 224 and for whom PK parameters could be adequately estimated. All participants included in the overall number of participants analyzed contributed data to this endpoint.
Measure: Mean (Full Range); unit: h*µg/mL
Arm/Group | Dose Exploration: AMG 224 Dose A | Dose Exploration: AMG 224 Dose B | Dose Exploration: AMG 224 Dose C | Dose Exploration: AMG 224 Dose D | Dose Exploration: AMG 224 Dose E | Dose Exploration: AMG 224 Dose F | Dose Exploration: AMG 224 Dose G | Dose Expansion: AMG 224 3 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 6 | 4 | 8
h*µg/mL
  AUC(3weeks): AMG 224 Conjugated Antibody after Cycle 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 2 | 8
  AUC(3weeks): AMG 224 Conjugated Antibody after Cycle 1 | 1850 [1240 to 2560] | 3450 [2870 to 4240] | 4520 [3910 to 4950] | 5260 [2750 to 7570] | 3710 [1590 to 4970] | 10400 [9040 to 14300] | 10500 [7060 to 14000] | 9690 [5620 to 14000]
  AUC(3weeks): AMG 224 Conjugated Antibody after Cycle 2: number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 3 | 1 | 7
  AUC(3weeks): AMG 224 Conjugated Antibody after Cycle 2 | 2330 [1340 to 2900] | 3650 [3460 to 3840] | 6360 [5820 to 7250] | 7400 [4000 to 9640] | 7610 [4250 to 12400] | 14100 [13100 to 15100] | 23000 [23000 to 23000] | 15500 [10100 to 20800]
  AUC(3weeks): Total Anti-BCMA Antibody after Cycle 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 2 | 8
  AUC(3weeks): Total Anti-BCMA Antibody after Cycle 1 | 1990 [1300 to 2690] | 3850 [3300 to 4450] | 5120 [4540 to 5910] | 5870 [3160 to 8110] | 4220 [2200 to 5440] | 11300 [10400 to 12500] | 11200 [6140 to 16200] | 8680 [6640 to 11400]
  AUC(3weeks): Total Anti-BCMA Antibody after Cycle 2: number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 3 | 1 | 7
  AUC(3weeks): Total Anti-BCMA Antibody after Cycle 2 | 2530 [1460 to 3310] | 4370 [4180 to 4560] | 8140 [7140 to 10100] | 9170 [4660 to 13200] | 9250 [4900 to 16100] | 18500 [17400 to 20500] | 24700 [24700 to 24700] | 13000 [8880 to 18600]
  AUC(0-96hr): DM1 after Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 5 | 3 | 4
  AUC(0-96hr): DM1 after Cycle 1 |  |  |  |  | 0.0729 [0.0729 to 0.0729] | 0.0487 [0.0328 to 0.0597] | 0.0579 [0.0421 to 0.0668] | 0.0646 [0.0426 to 0.0743]
  AUC(0-96hr): DM1 after Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 5 | 1 | 7
  AUC(0-96hr): DM1 after Cycle 2 |  |  |  |  | 0.0561 [0.0561 to 0.0561] | 0.0654 [0.0484 to 0.0770] | 0.0684 [0.0684 to 0.0684] | 0.0688 [0.0588 to 0.0865]

6. Secondary Outcome: Clearance (CL) of AMG 224 Conjugated Antibody, Total Anti-BCMA Antibody, and Total Unconjugated DM1
Description: CL of AMG 224 conjugated antibody, total anti-BCMA antibody and total unconjugated DM1 was determined.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Full Range); unit: mL/hr
Arm/Group | Dose Exploration: AMG 224 Dose A | Dose Exploration: AMG 224 Dose B | Dose Exploration: AMG 224 Dose C | Dose Exploration: AMG 224 Dose D | Dose Exploration: AMG 224 Dose E | Dose Exploration: AMG 224 Dose F | Dose Exploration: AMG 224 Dose G | Dose Expansion: AMG 224 3 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 6 | 5 | 10
mL/hr
  AMG 224 Conjugated Antibody after Cycle 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 10
  AMG 224 Conjugated Antibody after Cycle 1 | 17.7 [11.7 to 24.2] | 17.9 [14.2 to 20.9] | 20.1 [18.2 to 23.0] | 27.2 [15.8 to 43.7] | 47.0 [28.2 to 100] | 18.8 [13.3 to 21.0] | 26.0 [17.9 to 35.4] | 26.6 [15.1 to 42.7]
  AMG 224 Conjugated Antibody after Cycle 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 2 | 7
  AMG 224 Conjugated Antibody after Cycle 2 | 14.5 [10.3 to 22.3] | 15.9 [14.8 to 17.3] | 14.3 [12.4 to 15.5] | 18.8 [12.4 to 30.0] | 25.5 [12.9 to 37.7] | 13.7 [9.13 to 18.8] | 20.9 [10.9 to 30.9] | 16.1 [11.2 to 22.8]
  Total Anti-BCMA Antibody after Cycle 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 9
  Total Anti-BCMA Antibody after Cycle 1 | 16.5 [11.1 to 23.2] | 15.8 [13.5 to 18.2] | 17.8 [15.2 to 19.8] | 23.9 [14.8 to 38.0] | 40.5 [25.7 to 72.8] | 16.8 [15.2 to 18.3] | 24.6 [15.5 to 40.7] | 26.2 [12.9 to 34.6]
  Total Anti-BCMA Antibody after Cycle 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 2 | 8
  Total Anti-BCMA Antibody after Cycle 2 | 13.4 [9.07 to 20.5] | 13.4 [12.9 to 14.3] | 11.4 [8.92 to 12.6] | 15.8 [9.10 to 25.8] | 22.1 [9.94 to 32.6] | 11.4 [9.29 to 16.2] | 22.4 [10.1 to 34.6] | 18.6 [11.6 to 24.8]
  DM1 after Cycle 1: number analyzed (Participants) | 0 | 0 | 2 | 3 | 5 | 6 | 5 | 10
  DM1 after Cycle 1 |  |  | 20800000 [20400000 to 21300000] | 53300000 [6310000 to 131000000] | 9310000 [2190000 to 24300000] | 4360000 [3180000 to 5790000] | 6100000 [3740000 to 9350000] | 5620000 [2160000 to 10600000]
  DM1 after Cycle 2: number analyzed (Participants) | 0 | 1 | 3 | 3 | 2 | 5 | 2 | 7
  DM1 after Cycle 2 |  | 18700000 [18700000 to 18700000] | 69800000 [13500000 to 173000000] | 11300000 [5860000 to 21700000] | 5060000 [2850000 to 7270000] | 2990000 [2470000 to 3930000] | 5970000 [3660000 to 8290000] | 3480000 [2080000 to 4960000]

7. Secondary Outcome: Terminal Half-life (t1/2,z) of AMG 224 Conjugated Antibody, Total Anti-BCMA Antibody, and Total Unconjugated DM1
Description: The t1/2,z of AMG 224 conjugated antibody, total anti-BCMA antibody and total unconjugated DM1 was measured.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Exploration: AMG 224 Dose A | Dose Exploration: AMG 224 Dose B | Dose Exploration: AMG 224 Dose C | Dose Exploration: AMG 224 Dose D | Dose Exploration: AMG 224 Dose E | Dose Exploration: AMG 224 Dose F | Dose Exploration: AMG 224 Dose G | Dose Expansion: AMG 224 3 mg/kg
Number analyzed (Participants) | 3 | 3 | 1 | 2 | 5 | 1 | 2 | 6
hours
  AMG 224 Conjugated Antibody after Cycle 1: number analyzed (Participants) | 2 | 3 | 1 | 2 | 3 | 1 | 2 | 3
  AMG 224 Conjugated Antibody after Cycle 1 | 217 [217 to 218] | 218 [191 to 284] | 278 [278 to 278] | 196 [174 to 219] | 139 [135 to 160] | 189 [189 to 189] | 195 [192 to 198] | 199 [158 to 217]
  AMG 224 Conjugated Antibody after Cycle 2: number analyzed (Participants) | 3 | 2 | 0 | 2 | 3 | 1 | 1 | 3
  AMG 224 Conjugated Antibody after Cycle 2 | 201 [194 to 215] | 221 [193 to 249] |  | 189 [159 to 220] | 243 [155 to 300] | 164 [164 to 164] | 179 [179 to 179] | 241 [174 to 280]
  Total Anti-BCMA Antibody after Cycle 1: number analyzed (Participants) | 2 | 1 | 0 | 2 | 4 | 1 | 1 | 2
  Total Anti-BCMA Antibody after Cycle 1 | 234 [231 to 238] | 198 [198 to 198] |  | 242 [197 to 287] | 155 [51.0 to 189] | 238 [238 to 238] | 170 [170 to 170] | 194 [172 to 216]
  Total Anti-BCMA Antibody after Cycle 2: number analyzed (Participants) | 3 | 1 | 0 | 2 | 1 | 0 | 1 | 4
  Total Anti-BCMA Antibody after Cycle 2 | 269 [250 to 277] | 255 [255 to 255] |  | 230 [211 to 249] | 351 [351 to 351] |  | 147 [147 to 147] | 199 [157 to 290]
  DM1 after Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
  DM1 after Cycle 1 |  |  |  |  | 50.2 [50.2 to 50.2] | 52.1 [52.1 to 52.1] |  | 48.8 [48.8 to 48.8]
  DM1 after Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Best Overall Response (BOR) According to International Myeloma Working Group Uniform Response Criteria (IMWG-URC)
Description: BOR was the best observed post baseline disease response per IMWG-URC: Complete response (CR): Negative immunofixation on serum and urine, soft tissue plasmacytomas disappearance, < 5% plasma cells in bone marrow (BM). Stringent CR (sCR): CR and normal serum free light chain ratio and no clonal cells in BM. Very Good Partial Response (VGPR): Serum and urine M-protein detectable by immunofixation or ≥ 90% reduction in serum M-protein (urine M-protein level < 100 mg/24-h). PR: ≥ 50% reduction of serum M-protein and 24-h urinary M-protein by ≥ 90% or to < 200 mg/24-h. Minor Response (MR): 25-49% reduction of serum M-protein and 50-89% in 24-h urinary M-protein, exceeding 200 mg/24-h. Stable Disease (SD): Not meeting criteria for CR, VGPR, PR or Progressive Disease (PD). PD: ≥ 25% increase in serum or urine M-component, development of new or increased size of existing bone lesions or soft tissue plasmacytomas, hypercalcemia attributed to the plasma cell proliferative disorder.
Time Frame: Day 1 of Cycle 1 to up to the end of study visit; up to approximately 6 years
Population: Safety analysis set included all participants who received at least 1 dose of AMG 224.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Exploration: AMG 224 Dose A | Dose Exploration: AMG 224 Dose B | Dose Exploration: AMG 224 Dose C | Dose Exploration: AMG 224 Dose D | Dose Exploration: AMG 224 Dose E | Dose Exploration: AMG 224 Dose F | Dose Exploration: AMG 224 Dose G | Dose Expansion: AMG 224 Dose H + Prior CD38 Targeting Antibody Treatment | Dose Expansion: AMG 224 Dose H + no Prior CD38 Targeting Antibody Treatment
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 9 | 2
Participants
  sCR | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  VGPR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  PR | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
  MR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  SD | 2 | 1 | 1 | 2 | 1 | 2 | 1 | 2 | 0
  Progressive disease | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 0
  Unevaluable | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 2 | 1

9. Secondary Outcome: Time To Progression (TTP) According to IMWG-URC
Description: TTP was the time from the first administration of AMG 224 to the first objective assessment of disease progression as per IMWG-URC or deaths or if applicable date of censoring. The median TTP was estimated using the Kaplan-Meier method
Time Frame: Day 1 of Cycle 1 to up to the end of study visit; up to approximately 6 years
Population: The safety analysis set included all participants who received at least 1 dose of AMG 224.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Dose Exploration: AMG 224 Dose A | Dose Exploration: AMG 224 Dose B | Dose Exploration: AMG 224 Dose C | Dose Exploration: AMG 224 Dose D | Dose Exploration: AMG 224 Dose E | Dose Exploration: AMG 224 Dose F | Dose Exploration: AMG 224 Dose G | Dose Expansion: AMG 224 Dose H + Prior CD38 Targeting Antibody Treatment | Dose Expansion: AMG 224 Dose H + no Prior CD38 Targeting Antibody Treatment
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 9 | 2
months | 74.9 [3.5 to NA] — Too few events to estimate the upper 80% confidence interval (CI) | 1.6 [0.7 to NA] — Too few events to estimate the upper 80% CI | 1.4 [0.8 to NA] — Too few events to estimate the upper 80% CI | 3.7 [2.1 to NA] — Too few events to estimate the upper 80% CI | 14.0 [11.6 to NA] — Too few events to estimate the upper 80% CI | 2.3 [1.4 to 6.0] | 2.8 [0.7 to NA] — Too few events to estimate the upper 80% CI | 7.2 [0.7 to 12.3] | 4.4 [0.3 to NA] — Too few events to estimate the upper 80% CI

10. Secondary Outcome: Duration of Response (DOR) According to IMWG-URC
Description: DOR was defined as the time between the date of the first observation indicating an objective response as PR (or better) through to the subsequent date of disease progression as classified by the IMWG-URC for Multiple Myeloma or death or where applicable date of censoring. The median DOR was estimated using the Kaplan-Meier method.
Time Frame: Day 1 of Cycle 1 to up to the end of study visit; up to approximately 6 years
Population: The safety analysis set included all participants who received at least 1 dose of AMG 224.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Dose Exploration: AMG 224 Dose A | Dose Exploration: AMG 224 Dose B | Dose Exploration: AMG 224 Dose C | Dose Exploration: AMG 224 Dose D | Dose Exploration: AMG 224 Dose E | Dose Exploration: AMG 224 Dose F | Dose Exploration: AMG 224 Dose G | Dose Expansion: AMG 224 Dose H + Prior CD38 Targeting Antibody Treatment | Dose Expansion: AMG 224 Dose H + no Prior CD38 Targeting Antibody Treatment
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 9 | 2
months | 63.1 [NA to NA] — Too few events to estimate the 80% CIs | NA [NA to NA] — No events therefore median and 80% CIs could not be estimated | NA [NA to NA] — No events therefore median and 80% CIs could not be estimated | 60.8 [NA to NA] — Too few events to estimate the 80% CIs | 9.1 [8.1 to NA] — Too few events to estimate the upper 80% CI | 19.2 [NA to NA] — Too few events to estimate the 80% CIs | 4.1 [NA to NA] — Too few events to estimate the 80% CIs | 18.7 [6.7 to NA] — Too few events to estimate the upper 80% CI | 7.7 [NA to NA] — Too few events to estimate the 80% CIs

11. Secondary Outcome: Number of Participants With Conversion to Minimal Residual Disease (MRD)-Negativity
Description: MRD negative was defined as a tumor load of less than 1 clonal cell in 10^5 normal cells (as determined by flow cytometry).
Time Frame: Day 1 of Cycle 1 to up to the end of study visit; up to approximately 6 years
Population: Safety analysis set: all participants that are enrolled and received at least 1 dose of AMG 224.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Exploration: AMG 224 Dose A | Dose Exploration: AMG 224 Dose B | Dose Exploration: AMG 224 Dose C | Dose Exploration: AMG 224 Dose D | Dose Exploration: AMG 224 Dose E | Dose Exploration: AMG 224 Dose F | Dose Exploration: AMG 224 Dose G | Dose Expansion: AMG 224 Dose H + Prior CD38 Targeting Antibody Treatment | Dose Expansion: AMG 224 Dose H + no Prior CD38 Targeting Antibody Treatment
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 9 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Anti-AMG 224 Antibodies
Description: The number of participants who tested positive for pre-existing binding antibodies prior to exposure to AMG 224 and who tested positive for anti-AMG 224 binding antibodies after dosing with AMG 224 are presented. Participants with transient post-baseline results were binding antibody positive post-baseline with a negative or no result at baseline and a negative result at the participant's last timepoint tested.
Time Frame: Day 1 of Cycle 1 to up to the end of study visit; up to approximately 6 years
Population: The safety analysis set included all participants who received at least 1 dose of AMG 224.
Measure: Number; unit: participants
Arm/Group | Dose Exploration: AMG 224 Dose A | Dose Exploration: AMG 224 Dose B | Dose Exploration: AMG 224 Dose C | Dose Exploration: AMG 224 Dose D | Dose Exploration: AMG 224 Dose E | Dose Exploration: AMG 224 Dose F | Dose Exploration: AMG 224 Dose G | Dose Expansion: AMG 224 Dose H + Prior CD38 Targeting Antibody Treatment | Dose Expansion: AMG 224 Dose H + no Prior CD38 Targeting Antibody Treatment
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 9 | 2
participants
  Binding antibody positive at anytime | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1
  Binding antibody positive at/before baseline | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Binding antibody positive post-baseline with a negative/no result at baseline | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Binding antibody positive post-baseline with a negative/no result at baseline: Transient | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected from enrollment to the end of study visit, up to approximately 6 years. Treatment-emergent adverse events were collected from the first administration of AMG 224 up to 37 days after the last dose of investigational product (median treatment duration was 9 weeks).
Description: Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- Dose Exploration: AMG 224 Dose A: Participants were administered AMG 224 Dose A as an IV infusion Q3W on Day 1 of each cycle, where each cycle is 3 weeks.
Arm/Group | Dose Exploration: AMG 224 Dose A | Dose Exploration: AMG 224 Dose B | Dose Exploration: AMG 224 Dose C | Dose Exploration: AMG 224 Dose D | Dose Exploration: AMG 224 Dose E | Dose Exploration: AMG 224 Dose F | Dose Exploration: AMG 224 Dose G | Dose Expansion: AMG 224 Dose H + Prior CD38 Targeting Antibody Treatment | Dose Expansion: AMG 224 Dose H + no Prior CD38 Targeting Antibody Treatment
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/6 | 0/6 | 0/5 | 0/11 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 0/3 | 2/3 | 2/6 | 2/6 | 2/5 | 6/9 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 5/6 | 6/6 | 5/5 | 7/9 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Exploration: AMG 224 Dose A (N=3) | Dose Exploration: AMG 224 Dose B (N=3) | Dose Exploration: AMG 224 Dose C (N=3) | Dose Exploration: AMG 224 Dose D (N=3) | Dose Exploration: AMG 224 Dose E (N=6) | Dose Exploration: AMG 224 Dose F (N=6) | Dose Exploration: AMG 224 Dose G (N=5) | Dose Expansion: AMG 224 Dose H + Prior CD38 Targeting Antibody Treatment (N=9) | Dose Expansion: AMG 224 Dose H + no Prior CD38 Targeting Antibody Treatment (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Plasma cell disorder (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Exploration: AMG 224 Dose A (N=3) | Dose Exploration: AMG 224 Dose B (N=3) | Dose Exploration: AMG 224 Dose C (N=3) | Dose Exploration: AMG 224 Dose D (N=3) | Dose Exploration: AMG 224 Dose E (N=6) | Dose Exploration: AMG 224 Dose F (N=6) | Dose Exploration: AMG 224 Dose G (N=5) | Dose Expansion: AMG 224 Dose H + Prior CD38 Targeting Antibody Treatment (N=9) | Dose Expansion: AMG 224 Dose H + no Prior CD38 Targeting Antibody Treatment (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 3 | 5 | 3 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Splenic lesion (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 2 | 2 | 1 | 5 | 3 | 6 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 3 | 1 | 0 | 4 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 1 | 4 | 2 | 3 | 1
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 0 | 3 | 3 | 4 | 0 | 6 | 0
Infusion site bruising (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 2 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes ophthalmic (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 1 | 1 | 1 | 3 | 2 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 1 | 1 | 1 | 4 | 2 | 4 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 3 | 1
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Calcium ionised increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coagulation time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 2 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2 | 2 | 0 | 5 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 2 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin neoplasm excision (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Product after taste (Product Issues) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spider naevus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT02561962/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT02561962/SAP_001.pdf